CLINICAL TRIAL: NCT02793713
Title: Prospective Validation of a Malignancy Scoring System During Endoscopic Evaluation of Mediastinal Lymph Nodes for Lung Cancer
Brief Title: EBUS Score Validation for Malignancy
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Toronto General Hospital (Other); Vancouver General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EBUS_ScoreValidation
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Lung Neoplasms; Lung Diseases
Keywords: EBUS; Prediction; malignancy; lymph nodes; lung cancer; Diagnostic Techniques, Respiratory System
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endobronchial Ultrasound — Patients undergoing EBUS with TransBronchial Needle Aspiration will be invited to enroll on the day of their procedure. Once informed consent is obtained, the surgeon will assess the sonographic criteria, take pictures, and biopsy every lymph node of interest. All three elements of this assessment will need to be completed for a specimen to be included in the study. After the procedure, the operating surgeon will fill the Lymph Node Assessment questionnaire, assign an aggregate score to every lymph node specimen, and attach the pictures to the form. Pictures from every specimen will stored electronically to be reviewed and secondarily rated by a second blinded surgeon. Patient involvement in the study ends at the completion of the planned procedure.
  Other Names: EBUS

SUMMARY:
Surgical removal of a tumour in the lung offers the best chance for survival in early stage lung cancers. One main criteria of surgical eligibility is the absence of cancer spread to the lymph nodes; rendering the staging process extremely important. The evaluation of these lymph nodes is thought to be best completed using Endobronchial Ultrasound (EBUS), a procedure in which several lymph nodes are sampled and send to pathology to determine whether or not it is malignant. More recently, studies have observed that there are clear differences in the characteristics of cancerous and benign (non-cancerous) lymph nodes, and so there has been great interest in creating a list of criteria that can determine whether a node is malignant. This study aims to prospectively validate a previously proposed score based on observed characteristics of lymph nodes during an EBUS procedure relating to pathology-confirmed results. To test this, the results of the lymph node samples and the observed score will be compared for agreement. If the investigators find that the scoring system can accurately predict which lymph nodes are cancerous, it would provide the evidence to establish the score as a standard procedure during cancer staging.

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with confirmed or suspected lung cancer and be undergoing EBUS diagnosis/staging

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with suspected or confirmed NSCLC and have been referred to mediastinal staging via EBUS at St. Joseph's Healthcare Hamilton, Toronto General Hospital, Vancouver General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-06; Primary Completion 2017-09-17 (Actual); Study Completion 2017-09-17 (Actual)

PRIMARY OUTCOMES:
Internal validity of an aggregate sonographic score | Duration of EBUS procedure (estimated 1 hour)
  Objective is to compare the lymph node malignancy predictor score obtained by two raters, one who performed the procedure and the other a secondary rater who viewed the video of the procedure. The score will ideally be similar between raters, showing good inter-rater internal validity.
External validity of an aggregate sonographic score | From time of EBUS procedure to date of surgery (expected to be up to 1 month)
  As the gold standard for lymph node assessment is via tissue sampling obtained during an EBUS (or other invasive method) procedure, the scores obtained using the lymph node malignancy predictor scoring technique will be compared to later post-surgical pathological staging. The score will be considered to have good criterion (external) validity if there is a high degree of agreement between the pathology and score values.

SECONDARY OUTCOMES:
Rate of staging re-intervention after initial EBUS | Up to 12 months
  If the original tissue samples taken during the EBUS procedure were found to be insufficient to rule out malignancy, the patient may undergo another EBUS, or will undergo an Endoscopic ultrasound or a mediastinoscopy. During these follow-up procedures, the surgeon would be obtaining additional tissue in the hope that a result can be made. These re-intervention is not without a risk of adverse events, and ideally should be minimized. We will be abstracting re-intervention occurrences from patient charts.
Correlation between lymph node aggregate sonographic score and Positron Emission Tomography-elicited Standardized Uptake Values (SUVs) | From first presentation for diagnosis to date of surgery (Estimated to be 2-3 months)
  All patients undergo Positron Emission Tomography in the course of their clinical staging for suspected lung cancer. The values obtained from this diagnostic test (Standardized Uptake Values [SUVs]) will be obtained and compared to the surgeon's observed score on the lymph node aggregate sonographic scoring tool to investigate whether there is any relationship between the score and the SUVs.

CONTACTS AND LOCATIONS:
Overall Officials: Wael C Hanna, MDCM MBA, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Chest Physicians; Health and Science Policy Committee. Diagnosis and management of lung cancer: ACCP evidence-based guidelines. American College of Chest Physicians. Chest. 2003 Jan;123(1 Suppl):D-G, 1S-337S. No abstract available. PMID 12527560
- [Background] Hanna WC, Yasufuku K. Bronchoscopic staging of lung cancer. Ther Adv Respir Dis. 2013 Apr;7(2):111-8. doi: 10.1177/1753465812468041. Epub 2012 Dec 20. PMID 23258501
- [Background] Schmid-Bindert G, Jiang H, Kahler G, Saur J, Henzler T, Wang H, Ren S, Zhou C, Pilz LR. Predicting malignancy in mediastinal lymph nodes by endobronchial ultrasound: a new ultrasound scoring system. Respirology. 2012 Nov;17(8):1190-8. doi: 10.1111/j.1440-1843.2012.02223.x. PMID 22789110
- [Background] Shafiek H, Fiorentino F, Peralta AD, Serra E, Esteban B, Martinez R, Noguera MA, Moyano P, Sala E, Sauleda J, Cosio BG. Real-time prediction of mediastinal lymph node malignancy by endobronchial ultrasound. Arch Bronconeumol. 2014 Jun;50(6):228-34. doi: 10.1016/j.arbres.2013.12.002. Epub 2014 Feb 8. English, Spanish. PMID 24512940
- [Background] Wang L, Wu W, Hu Y, Teng J, Zhong R, Han B, Sun J. Sonographic Features of Endobronchial Ultrasonography Predict Intrathoracic Lymph Node Metastasis in Lung Cancer Patients. Ann Thorac Surg. 2015 Oct;100(4):1203-9. doi: 10.1016/j.athoracsur.2015.04.143. Epub 2015 Jul 28. PMID 26228606
- [Background] El-Sherief AH, Lau CT, Wu CC, Drake RL, Abbott GF, Rice TW. International association for the study of lung cancer (IASLC) lymph node map: radiologic review with CT illustration. Radiographics. 2014 Oct;34(6):1680-91. doi: 10.1148/rg.346130097. PMID 25310423